CLINICAL TRIAL: NCT07373028
Title: A Randomized Controlled Trial to Explore the Long-term Effects of a Simple Swallowing Training Program on Older Individuals in the Community
Brief Title: Simple Swallowing Training Program on Older Individuals in the Community
Acronym: SSTP1year
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zeng Changhao (Other)
Responsible Party: Sponsor-Investigator, Zeng Changhao, Principle Investigator, People's Hospital of Zhengzhou University
Organization: People's Hospital of Zhengzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SSTPlongterm
Record Dates: First submitted 2026-01-12; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Dysphagia
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simple swallowing training program group (Experimental): Older individuals will be assigned to the simple swallowing training program, with rest on weekends, and training conducted only on weekdays, twice a day for 15 minutes each time. Each training session will take place approximately one hour before meals. Online guidance services will be provided by the researchers.
  Interventions: Behavioral: Simple swallowing training program
- Active control group (Active Comparator): Participants in the active control group are assigned to physical activities that correspond to the amount, frequency, and duration of the simple swallowing training program. These activities are designed to minimize any impact on swallowing function while being considered sufficient to reduce the potential effects associated with physical activity. Online guidance services will be provided by the researchers.
  Interventions: Behavioral: Active non-swallowing training

INTERVENTIONS:
Behavioral: Simple swallowing training program — The Simple swallowing training program included warm-up and another 11 sections, including Warm-up for 3 min, Neck Activation for 1 min, Nod for 1 min, Lip Closure for 1 min, Cheek Puffing for 1 min, Breathing Exercise for 1 min, Voice Training for 2 min, Swallowing Exercise for 2-3 min, Neck Massage for 1 min, Acupressure for 2 min, Facial Massage for 3 min and Tongue Exercise for 1 min.
  Arms: Simple swallowing training program group
Behavioral: Active non-swallowing training — A set of light physical activities that will not affect swallowing function, lasting approximately 15 minutes, similar to the simple swallowing training program and requiring no equipment.
  Arms: Active control group

SUMMARY:
The goal of this clinical trial is to explore the effects of a simple swallowing training program on the swallowing function, airway protection, nutritional risk, daily choking, quality of life, and mental health of elderly individuals with mild swallowing difficulties residing in the community. The main question it aims to answer is: Does the simple swallowing training program significantly improve participants' swallowing function and safety, as well as their quality of life? Additionally, can daily choking incidents be improved?

DETAILED DESCRIPTION:
The goal of this clinical trial is to explore the effects of a simple swallowing training program on the swallowing function, airway protection, nutritional risk, daily choking, quality of life, and mental health of elderly individuals with mild swallowing difficulties residing in the community. The main question it aims to answer is: Does the simple swallowing training program significantly improve participants' swallowing function and safety, as well as their quality of life? Additionally, can daily choking incidents be improved? Additionally, the investigator will compare the long-term effects of the training with the previous study to see the significance of long-term training.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 years or older and living in communities.
* Speaking Chinese
* Daily oral feeding.
* The swallowing risk was detected through the Volume-Viscosity Swallow Test, and mild dysphagia based on Dysphagia Outcome and Severity Scale
* No history of hospitalization in the past 6 months.
* No participation in any swallowing-related intervention in the past 6 months.
* Conscious and able to cooperate with questionnaires and training.

Exclusion Criteria:

* Self-reported medical condition precluding exercise.
* Physical disability.
* Abnormalities of the oral, pharyngeal, or esophageal structures.
* Diagnosis of aspiration pneumonia.
* Presence of a tracheostomy
* Neuromuscular disorders
* Cognitive impairment

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 474 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Dysphagia Outcome and Severity Scale | day 0 and day 366
  The Dysphagia Outcome and Severity Scale consists of 7 levels, from 1 to 7, based on imaging data. A higher level indicates better swallowing function.

SECONDARY OUTCOMES:
Aspiratory cough | 1 year
  Aspiratory cough is based on self-reporting and recorded via paper or electronic calendars, which are periodically uploaded. Cough is defined as the coughing and discomfort caused by food or water entering the airway for various reasons. The outcomes of choking include relief through actions such as coughing or patting the back, or no relief at all.
Nutrition Risk Screening 2002 | day 0, day 183 and day 366
  Nutrition Risk Screening 2002 is a tool used to assess nutritional risk. The total score ranges from 0 to 7, with a score of 3 or higher indicating the presence of nutritional risk.
Dysphagia Handicap Index | day 0, day 31, day 183 and day 366
  Dysphagia Handicap Index is used to assess quality of life. The total score ranges from 0 to 100, with the higher score indicating worse quality of life.
Penetration-Aspiration Scale | day 0 and day 366
  Penetration-Aspiration Scale is used to assess airway protection. The total score ranges from 1 to 8, with the higher score indicating worse airway protection.
Aspiration pneumonia | 1 year
  Participants are monitored for the occurrence of aspiration pneumonia, with the standard being the diagnosis issued by the hospital. It is considered that a participant may experience aspiration pneumonia multiple times within a year. Based on imaging results, aspiration pneumonia resulting from the same incident of aspiration is regarded as the same positive case. Participants or their relatives are required to regularly submit information regarding their pneumonia.
10-item Eating assessment tool | day 0, day 31, day 183 and day 366
  10-item Eating assessment tool was used to assess subject swallowing ability. The total score ranges from 0 to 40, with the higher score indicating more severe subject swallowing disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Xi Zeng, PhD, Study Director — ZZU First Hospital
Locations (2):
- China (2):
  - Gaoxin Qu, Suzhou
  - Huiji Jinshui Gaoxin Erqi Qu, Zhenzhou